CLINICAL TRIAL: NCT06850155
Title: Impact of Gluteal Sling Release on Gluteal Dysfunction and Functional Outcomes in Primary Total Hip Arthroplasty
Brief Title: Gluteal Sling Release on Gluteal Dysfunction After in Primary Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Enejd Veizi, MD, MD, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-23-4913
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hip Osteoarthritis; Osteoarthritis, Hip; Gluteus Maximus Muscle Atrophy; Muscle Weakness Condition; Fatty Degeneration
Keywords: hip arthroplasty; gluteal sling; muscle atrophy; gluteus maximus
MeSH Terms: conditions — Osteoarthritis, Hip; Fatty Liver; Muscular Atrophy | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Gluteal Sling (No Intervention): The Gluteal sling was left untouched during the whole procedure
- Released Gluteal Sling (Experimental): The Gluteal sling was released and left unrepaired at the end of the procedure
  Interventions: Procedure: Sling release
- Released&Repaired Gluteal Sling (Experimental): The Gluteal sling was released and then repaired at the end of the procedure
  Interventions: Procedure: Sling release and repair

INTERVENTIONS:
Procedure: Sling release — The gluteal sling was released and left unrepaired at the end of the procedure
  Arms: Released Gluteal Sling
Procedure: Sling release and repair — The gluteal sling was released and then repaired at the end of the procedure
  Arms: Released&Repaired Gluteal Sling

SUMMARY:
This study investigates the effects of gluteal sling release during total hip arthroplasty (THA) on gluteal muscle function and hip joint performance. The gluteal sling release technique is used to improve surgical visualization and reduce the risk of sciatic nerve compression, but its impact on postoperative muscle function remains unclear. A prospective randomized controlled trial was conducted on 144 patients with unilateral coxarthrosis undergoing THA, divided into three groups: gluteal sling preserved, released, and released with repair. Clinical outcomes were assessed preoperatively and at six months postoperatively using VAS, HHS, and WOMAC scores, alongside hip CT scans and isokinetic strength testing. While all groups showed significant functional improvement, muscle density in the released gluteal sling group decreased significantly, suggesting potential fatty degeneration. However, no significant differences were found in gluteus maximus surface area or hip extensor strength between the groups. The findings suggest that while gluteal sling release enhances intraoperative visualization and may reduce sciatic nerve injury risk, it could contribute to muscle degeneration. Therefore, preserving or repairing the sling when possible and implementing structured rehabilitation may optimize postoperative outcomes.

DETAILED DESCRIPTION:
This study aimed to assess the impact of gluteal sling release during total hip arthroplasty (THA) on gluteal muscle function and hip joint outcomes. A prospective randomized controlled trial was conducted between September 2023 and August 2024, including 144 patients diagnosed with unilateral coxarthrosis who underwent THA. Patients were divided into three groups: gluteal sling preserved (n=47), released (n=52), and released and repaired (n=45). Preoperative and postoperative evaluations at six months included clinical scoring (VAS, HHS, and WOMAC), hip computed tomography (CT) scans for muscle cross-sectional area and density, and isokinetic testing to measure hip extensor strength. Surgical and rehabilitative procedures were standardized across all groups, with a focus on evaluating the functional and radiological effects of gluteal sling release.

The results demonstrated that all groups experienced significant postoperative improvements in pain scores (VAS), hip function (HHS), and joint-related disability (WOMAC) (p<0.001). No significant differences were observed between the groups in terms of gluteus maximus muscle cross-sectional area (p>0.05). However, muscle density significantly decreased in the gluteal sling release group (p=0.022), suggesting fatty degeneration, while no significant changes were observed in the other groups. Hip extensor strength showed a decline in the gluteal sling release group and an increase in the other groups, but these differences were not statistically significant (p>0.05). Sciatic nerve injury was recorded in one patient (2.1%) from the preserved group but was absent in the other groups. No significant differences were found in sciatic nerve injury rates across the groups.

In conclusion, the gluteal sling release technique provides better intraoperative visualization and may reduce the risk of iatrogenic sciatic nerve injury by alleviating nerve compression. However, while it does not significantly affect hip extensor strength, it may contribute to muscle fatty degeneration. Given these findings, preserving or repairing the gluteal sling whenever feasible is recommended. Additionally, a well-structured rehabilitation program following surgery is crucial to optimize patient recovery and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unilateral coxarthrosis
* Scheduled for primary total hip arthroplasty (THA)
* Age between 18 and 90 years

Exclusion Criteria:

* Coxarthrosis secondary to:

  * Developmental hip dysplasia
  * Fracture-related pathology
* Conditions requiring revision surgery, including:

  * Periprosthetic fractures
  * Current or previous hip joint infections
  * Rotational or malalignment issues requiring revision
* Neuromuscular diseases
* History of prior hip surgeries, such as:

  * Hip arthroscopy
  * Core decompression
* Mobility-limiting conditions in the contralateral hip (e.g., osteoarthritis)
* Patients lost to follow-up or with incomplete data
* Patients who developed complications (e.g., infection, dislocation) within six months of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Muscle atrophy | Preoperative & Postoperative 6th month
  Muscle atrophy through cross-sectional area measurement on CT scans (number, cm^2)
Muscle density | Preoperative & Postoperative 6th month
  Muscle density measurements on CT scans (Hounsfield units - HU)
Kinematic assesment | Postoperative 6th month
  Muscle strength through kinematic assesment (Nm)

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Preoperative & Postoperative 6th month
  minimum value:0, maximum value 10, higher values mean worse outcome
Harris Hip Score (HHS) | Preoperative & Postoperative 6th month
  minimum value:0, maximum value 100, higher values mean better outcome
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Preoperative & Postoperative 6th month
  minimum value:0, maximum value 100, higher values mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Enejd Veizi, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be publicly shared but the data will be made available upon request.

REFERENCES:
- [Result] Imren Y, Karslioglu B, Dedeoglu SS, Cabuk H, Atar S, Gurbuz S, Gurbuz H. The effect of gluteus maximus tenotomy in primary total hip arthroplasty with posterior approach: Kinematic analysis of hip extensor strength. J Orthop Surg (Hong Kong). 2021 Jan-Apr;29(1):23094990211003349. doi: 10.1177/23094990211003349. PMID 33779410
- [Result] Uemura K, Takao M, Sakai T, Nishii T, Sugano N. Volume Increases of the Gluteus Maximus, Gluteus Medius, and Thigh Muscles After Hip Arthroplasty. J Arthroplasty. 2016 Apr;31(4):906-912.e1. doi: 10.1016/j.arth.2015.10.036. Epub 2015 Nov 10. PMID 26652475
- [Result] Homma D, Minato I, Imai N, Miyasaka D, Sakai Y, Horigome Y, Suzuki H, Dohmae Y, Endo N. Investigation on the measurement sites of the cross-sectional areas of the gluteus maximus and gluteus medius. Surg Radiol Anat. 2019 Jan;41(1):109-115. doi: 10.1007/s00276-018-2099-9. Epub 2018 Sep 6. PMID 30191287